**Protocol Number: ADCT-402-101** 

Official Title: Phase 1 Dose-escalation Study to Evaluate the Tolerability, Safety,

Pharmacokinetics, and Antitumor Activity of ADCT-402 in Patients with

Relapsed or Refractory B-cell Lineage Non Hodgkin Lymphoma (B-NHL)

NCT Number: NCT02669017

**Document Date: 10 June 2019** 

# **Statistical Analysis Plan**

A Phase 1 Dose-escalation Study to Evaluate the Tolerability, Safety, Pharmacokinetics, and Antitumor Activity of ADCT-402 in Patients with Relapsed or Refractory B-cell Lineage Non-Hodgkin Lymphoma (B-NHL)

PROTOCOL NO.: ADCT-402-101

**SAP Version No./ Date: 1.0/ Jun 10, 2019** 

Statistician: Luqiang Wang

## **Confidentiality Statement**

All financial and nonfinancial support for this study will be provided by ADC Therapeutics SA. The concepts and information contained in this document or generated during the study are considered proprietary and may not be disclosed in whole or in part without the expressed, written consent of ADC Therapeutics SA. The study will be conducted according to the International Conference on Harmonisation harmonised tripartite guideline E6(R1), Good Clinical Practice.

Signature

# SAP Approval – Sponsor Signatory

| Study Title | A Phase 1 Dose-escalation Study to Evaluate the Tolerability,<br>Safety, Pharmacokinetics, and Antitumor Activity of ADCT-<br>402 in patients with Relapsed or Refractory B-cell Lineage<br>Non-Hodgkin Lymphoma (B-NHL) |
|---|---|
| Protocol Number | ADCT-402-101 |
| Original SAP Version Date: | 10 Jun 2019 |
| SAP accepted and approved b David Ungar, MD Head of US Oncology Clinica ADC Therapeutics Signature | |
| Shui He, PhD Head of Biometrics ADC Therapeutics | June 13, 2019 |

Date

ADCT-402

# **Table of Contents**

| Ta | ble of Contents | 3 |
|---|---|---|
| 1 l | Introduction | 5 |
| 2 5 | Study Objectives | 6 |
| | 2.1 Primary Objectives | 6 |
| | 2.2 Secondary Objectives | |
| 3 5 | Study Design | 7 |
| | 3.1 Sample Size Consideration | 7 |
| | 3.2 Randomization | 7 |
| | 3.3 Modifications to the statistical section of the protocol | 7 |
| 4 5 | Statistical methods | |
| | 4.1 Analysis Sets | 8 |
| | 4.1.1 Safety Analysis Set | |
| | 4.1.2 DLT-evaluable Analysis Set (Part 1) | |
| | 4.1.3 Efficacy Analysis Set | |
| | 4.1.4 Pharmacokinetics Analysis Set | 8 |
| | 4.2 Patient Disposition. | |
| | 4.3 Protocol Deviations | |
| | 4.4 Demographic and Baseline Characteristics | |
| | 4.5 Cancer History and Medications History | 10 |
| | 4.6 Prior or Concomitant Medications (other than anticancer therapies) | 11 |
| | 4.7 Exposure to Treatment | 11 |
| | 4.7.1 Extent of ADCT-402 Exposure | 11 |
| | 4.7.2 Prophylactic Medications for Hypersensitivity | 12 |
| | 4.7.3 Subsequent Anticancer Therapy or Procedure | 12 |
| | 4.8 Safety Analyses | 12 |
| | 4.8.1 Dose-limiting Toxicities (Part 1) | 12 |
| | 4.8.2 Adverse Events, Serious Adverse Events, and Deaths | 12 |
| | 4.8.2.1 Analyses of adverse events | 12 |
| | 4.8.2.2 Deaths | 14 |
| | 4.8.3 Laboratory Data | 14 |

| ADC Therapeutics | ADCT-402 |
|------------------------------------------------|-----------------|
| ADCT-402-101 | SAP version 1.0 |
| 4.8.4 Electrocardiogram | 15 |
| 4.8.5 Vital Signs | 15 |
| 4.8.6 ECOG Performance Status | 15 |
| 4.8.7 Physical Examinations and Body Weight | 15 |
| 4.9 Efficacy Analyses | 16 |
| 4.9.1 Overall Response Rate | 16 |
| 4.9.2 Duration of Response | 16 |
| 4.9.3 Time to Response: | 17 |
| 4.9.4 Progression-free Survival | 17 |
| 4.9.5 Overall Survival | 17 |
| 4.10 Pharmacokinetic/Pharmacodynamics Analyses | 18 |
| 4.10.1 PK Analysis Method | 18 |
| 5 Interim Analyses | |
| 6 Data handling conventions | 20 |
| 6.1 General conventions | 20 |
| 6.1.1 Missing data | 20 |
| 6.1.2 Unscheduled visits | 21 |
| 6.1.3 Duplicated visits | 21 |
| Appendix 1 Glossary of Abbreviations | 22 |

## 1 Introduction

This statistical analysis plan (SAP) describes the statistical methods to be used during the reporting and analyses of data collected under ADC Therapeutics Protocol ADCT-402-101.

This SAP should be read in conjunction with the study protocol and case report form (CRF). This version of the plan has been developed using the protocol Amendment 7 dated 16 October 2017 and CRF version 5 dated 23 Jan 2018.

## 2 Study Objectives

## 2.1 Primary Objectives

• Evaluate the safety and tolerability, and determine, as appropriate, the maximum tolerated dose (MTD) of ADCT-402 in patients with relapsed or refractory B-cell lineage NHL in Part 1.

- Determine the recommended dose(s) of ADCT-402 for Part 2 (expansion).
- Evaluate the safety and tolerability of ADCT-402 in Part 2 (expansion) at the dose level(s) recommended in Part 1.

## 2.2 Secondary Objectives

- Evaluate the clinical activity of ADCT-402 measured by overall response rate (ORR), duration of response (DOR), overall survival (OS), and progression-free survival (PFS).
- Characterize the pharmacokinetic (PK) profile of ADCT-402 (total antibody; drug-to-antibody ratio [DAR] ≥0), pyrrolobenzodiazepine (PBD)-conjugated antibody (DAR ≥ 1), and free warhead SG3199.
- Evaluate anti-drug antibodies (ADAs) to ADCT-402 in blood before, during, and after treatment with ADCT-402.



ADCT-402

ADCT-402

ADCT-402-101 SAP version 1.0

## 3 Study Design

This is a Phase 1, open-label, dose escalation (Part 1) and expansion (Part 2) study of the safety and tolerability of ADCT-402, used as monotherapy, in patients with relapsed or refractory B-cell NHL. The study will determine the MTD, as well as evaluate the preliminary activity, PK, pharmacodynamics (PD), and other exploratory assessments of ADCT-402.

In Part 1, patients will be assigned to treatment according to a 3+3 dose escalation design and oversight of a Dose Escalation Steering Committee (DESC). The initial dose of ADCT-402 will be 15  $\mu$ g/kg (Dose Level 1), and the highest allowed dose will be 300  $\mu$ g/kg. The dose-limiting toxicity (DLT) observation period for dose escalation is 1 cycle. Patients will be entered sequentially to each dose level. No intra-patient dose escalation is allowed. During Part 1, the DESC may expand enrollment at any dose level in which 3 patients have completed the DLT observation period if at least 1 patient in the study has achieved a partial response (PR) or better, or if further evaluation of PK or PD data is deemed necessary to characterize pharmacology in humans. No more than 10 patients in total can be treated at any dose level unless  $\geq$ 3 of the 10 patients have achieved a PR or better.

In Part 2, (expansion), all patients will be assigned to the dose level(s) of ADCT-402 identified in Part 1. During dose expansion, patients will be monitored for safety using the same DLT criteria employed during dose-escalation. If during the treatment period, >30% of patients experience safety events that would meet the criteria that define a DLT in the dose-escalation phase of the study, enrollment in the expansion cohort(s) may be paused and the study data reviewed to determine whether additional monitoring or other action (such as alternate dose levels) should be evaluated prior to further enrollment.

# 3.1 Sample Size Consideration

This is a Phase 1 study with a maximum sample size of up to approximately 200 patients. It is estimated that approximately 90 patients will enroll in Part 1, and approximately 110 patients will enroll in Part 2.

#### 3.2 Randomization

This study is not randomized.

# 3.3 Modifications to the statistical section of the protocol

The efficacy analysis set was defined in the protocol as all patients with valid baseline data who receive at least 2 doses of study drug or who have documented progression of disease at any time after the first dose of study drug. However, a few patients received 200  $\mu$ g/kg on an every 6 weeks (Q6W) schedule and their disease assessments were performed before the second dose. These patients should be considered as evaluable for efficacy analysis. Therefore, the efficacy analysis set is updated in the SAP to include all patients who have received at least one dose of ADCT-402 with a valid baseline and at least one valid post-baseline disease assessment or patients who have documented progression of disease or death at any time after the first dose of study drug.

#### 4 Statistical methods

All analyses use SAS® version 9.4 or higher. Summary tables will be organized by each dose level; if some dose levels have few patients, then dose levels could be combined into dose ranges. All available data will be used in the analyses, and important data will be included in data listings, sorted by dose level, patient, and by visit within patient. Missing data will not be imputed, except via censoring in survival analyses and as otherwise specified.

Unless otherwise noted, categorical data will be presented using counts and percentages, with the number of patients in the analysis set by treatment group as the denominator for percentages. Percentages will be rounded to one decimal place, except 100% will be displayed without any decimal places and percentages will not be displayed for zero counts. Continuous data, unless otherwise noted, will be summarized using the number of observations (n), mean, standard deviation (std), median, minimum, and maximum. Minima and maxima will be rounded to the precision of the original value, and means, medians, and 95% confidence intervals (CIs) if presented will be rounded to 1 decimal place greater than the precision of the original value. The std will be rounded to 2 decimal places greater than the precision of the original value, up to a maximum of 3 decimal places.

No hypothesis testing will be performed in this study.

#### 4.1 Analysis Sets

### 4.1.1 Safety Analysis Set

The safety analysis set consists of all patients who receive ADCT-402.

# 4.1.2 DLT-evaluable Analysis Set (Part 1)

The DLT-evaluable analysis set consists of patients who complete one cycle of ADCT-402. The patients with completed DLT information will be included even if they discontinue early, before the end of cycle 1.

# 4.1.3 Efficacy Analysis Set

The efficacy analysis set consists of patients who receive at least one dose of ADCT-402 with a valid baseline and at least one valid post-baseline disease assessment or patients who have documented progression of disease or death at any time after the first dose of study drug and before the start of any subsequent anticancer therapy or procedure.

# 4.1.4 Pharmacokinetics Analysis Set

The PK analysis set includes all patients who receive at least 1 dose of ADCT-402 with evaluable and sufficient concentration-time data to permit reliable estimation of ADCT-402 exposure, and with no major or critical protocol deviations related to ADCT-402 administration.



## **4.2 Patient Disposition**

The number and percentage of patients enrolled and treated in the study will be presented along with the number and percentage of patients in each analysis set for each dose level. In addition, for the safety analysis set, the number and percentage of patients who withdrew from study treatment and who discontinued the study for each reason will be tabulated for each dose level.

Patient disposition data will be listed.

#### 4.3 Protocol Deviations

The number and percentage of patients with any important clinical study report (CSR) reportable protocol deviation will be summarized overall and by type of deviation. The predefined important CSR reportable protocol deviations are listed below; in addition, any other protocol deviations deemed by ADCT medical to be important CSR reportable deviations will be included in the summary.

- 1. Patient entered the study even though they did not satisfy the entry criteria
- 2. Patient received a prohibited concomitant treatment during the study
- 3. Patients who met criteria for mandatory withdrawal of study drug during the study but did not have study drug withdrawn. The criteria for mandatory withdrawal of study drug included:
  - -Any patient who experiences a Grade 3 or higher hypersensitivity (Appendix 12.3 in the protocol) reaction, regardless of premedication, during any cycle of treatment.
  - -Any patient who experiences a recurrent Grade 3 or 4 toxicity, excluding hematological toxicity.
  - -Any patient who requires a dosing delay >21 consecutive days from the planned Day 1 dosing at any time during treatment (except in case of potential patient benefit, which must be approved by the Sponsor).

ADCT-402-101 SAP version 1.0

4. Patient who received the wrong treatment or incorrect dose. For example,

- -Actual dose of study drug was more than 15% greater than protocol defined planned dose level.
- -Patient started next cycle less than 18 days later after Day 1 of the most recent treatment cycle.

Important protocol deviations will be listed.

## 4.4 Demographic and Baseline Characteristics

Demographic and baseline characteristics will be tabulated for the safety analysis set by dose level. Variables include the following:

- Sex (female, male)
- Race (white, black or African American, Asian, American Indian or Alaska native, native Hawaiian or other Pacific Islander, other)
- Ethnicity (Hispanic or Latino, not Hispanic or Latino)
- Age (years)
- Age group ( $< 65, \ge 65 < 75, \ge 75 \text{ years}$ )
- Height (cm)
- Weight (kg)
- Body mass index (kg/m<sup>2</sup>)
- Eastern Cooperative Oncology Group (ECOG) performance status

Demographic and baseline characteristics data will be listed.

# 4.5 Cancer History and Medications History

Cancer history will be presented for the safety analysis set by dose level. Cancer history will include the following variables:

- Duration since diagnosis
- non-Hodgkin lymphoma subtype (diffuse large B-cell lymphoma, follicular lymphoma, chronic lymphocytic leukemia, mantle cell lymphoma, marginal zone B-cell lymphoma, Burkitt's lymphoma, lymphoplasmacytic lymphoma [Waldenstrom macroglobulinemia], other)
- Stage of disease (Stage I, II, III, IV; constitutional symptoms A, B; Subtype E, X, S)
- Cytogenetic analysis (results available yes, t(11;14), t(11q), +12, del(11q), del(13q), del(17p], t(14;18), t(8;14), t(8;22), other)
- Immunophenotypic analysis (results available yes; IgVH status mutated, unmutated, not applicable; CD5, CD10, CD19, CD20, CD21, CD23, CD43, CD79b, BCL1, BCL2, BCL6, CYCLIN D1, ZAP70 negative, positive, not done)

Prior anticancer procedure or therapy will include the following variables:

- Number of lines of therapy/ regimens per patient
- Any prior radiotherapy for the current malignancy (yes, no)
- Any prior systemic therapy for the current malignancy (yes, no)
- Reason for stopping therapy (progression, toxicity, other)

ADCT-402-101 SAP version 1.0

• Best response (complete response [CR], partial response [PR], stable disease [SD], progressive disease [PD], not evaluable [NE])

- Any prior stem cell transplant (yes, no)
- Type of transplant (allogenic, autologous, both, other)
- Conditioning therapy (yes, no)

Medical and cancer history data will be listed.

Prior anticancer radiotherapy, systemic therapy, and stem cell transplant data will be listed.

### 4.6 Prior or Concomitant Medications (other than anticancer therapies)

All medications taken within 14 days before dosing and until the end of the study are to be reported in the CRF pages.

All medications will be coded using the World Health Organization-Drug Dictionary (WHO-DD) and presented by dose level for the safety analysis set.

- Prior medications are those the patient used prior to first investigational product (IP) intake. Prior medications can be discontinued before first dosing or can be ongoing during the treatment phase.
- Concomitant medications are any treatments received by the patient concomitantly to any IP(s), from first dose (or start of the observation period) to the last dose + 30 days. A given medication can be classified both as a prior medication and as a concomitant medication. Concomitant medications do not include medications started 30 days after the last dose.

Any technical details related to computation, dates, and imputation for missing dates are described in Section 6.

Prior medications will be listed together with concomitant medications.

#### **4.7 Exposure to Treatment**

# 4.7.1 Extent of ADCT-402 Exposure

ADCT-402 exposure will be summarized for the safety analysis set by dose level. Duration of treatment, total number of cycles dosed, total dose received (in  $\mu g$  and  $\mu g/kg$ ), and average dose per cycle (in  $\mu g$  and  $\mu g/kg$ ) will be tabulated. When actual weight adjusted dose is needed, the last available weight before each infusion will be used. Dose administered at each infusion ( $\mu g$ ) is calculated by concentrated IP volume (in mL)\* 5 mg/mL \*1000 or serially diluted IP volume (in mL)/50\* 5 mg/mL \*1000; for partial infusion, multiply by (1-volume of dosing solution not administered [in mL]/ 50 mL).

Dose delays and dose reductions could also be analyzed if relevant. A cycle is delayed if it starts more than 3 days post-scheduled date.

Exposure data and infusion details will be listed together.

## 4.7.2 Prophylactic Medications for Hypersensitivity

Prophylactic medications for hypersensitivity will be listed only.

## 4.7.3 Subsequent Anticancer Therapy or Procedure

Patients' subsequent anticancer therapies or procedures including systemic therapy, radiation, transplant, or other, along with the start date of new anticancer therapy or procedure will be collected and listed only.

## 4.8 Safety Analyses

The summary of safety results will be presented by treatment group.

#### **General common rules**

All safety analyses will be performed on the safety analysis set, unless otherwise specified, using the following common rules:

- The baseline value is defined as the last non-missing value or measurement taken up to the first dose in the study.
- The analyses of the safety variables will be essentially descriptive and no systematic testing is planned.
- If relevant, selected safety analyses will be summarized by age, sex, racial subgroups, and any pertinent subgroups.
- The toxicity grade according to the Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 will be taken into account in the summary. For patients with multiple occurrences of the same event, the maximum grade is used. If a patient has both missing and non-missing severity grades for treatment-emergent adverse events (TEAEs) within the same preferred term (PT), the patient will be counted under the non-missing severity grade.

# **4.8.1 Dose-limiting Toxicities (Part 1)**

DLT data will be listed for Part 1 of the study.

## 4.8.2 Adverse Events, Serious Adverse Events, and Deaths

# 4.8.2.1 Analyses of adverse events

The primary focus of adverse event reporting will be on TEAEs. An adverse event (AE) will be considered to be a TEAE if it begins or worsens on or after first dose date and until 84 days (12 weeks) after the last dose date, or start of a new anticancer therapy/procedure, whichever comes earlier.

An AE occurring before the first dose or more than 84 days (12 weeks) after last dose date or after the start of a new anticancer therapy/procedure will not be included in TEAE displays, but will be listed as non-TEAEs.

ADCT-402-101 SAP version 1.0

If an AE date/time of onset (occurrence, worsening, or becoming serious) is incomplete, an imputation algorithm will be used to classify the AE as pre-treatment, TEAE, or post-treatment. The algorithm for imputing date/time of onset will be conservative and will classify an AE as a treatment-emergent unless there is definitive information to determine it is a non-TEAE (pre-or post-treatment).

Details on classification of AEs with missing or partial onset dates are provided in Section 6.

#### **Analysis of all TEAE(s):**

The following TEAE summaries will be generated for the safety analysis set in each dose level.

- Overview of TEAEs, summarizing number of TEAE and number (%) of patients with any
  - TEAE
  - Related TEAE (including possibly related, probably related, or related)
  - Any TEAE ≥Grade 3
  - Serious TEAE
  - TEAE leading to death
  - TEAE leading to permanent treatment withdrawal
  - TEAE leading to ADCT-402 delay or reduction
  - TEAE with at least one infusion related reaction
- All TEAEs \(\geq\)Grade 3 by PT, showing number (%) of patients with at least one TEAE, sorted by decreasing incidence of PTs
- All TEAEs by primary System Organ Class (SOC) and PT, showing number (%) of patients with at least one TEAE, sorted by SOC in alphabetic agreed order and decreasing incidence of PTs within SOC. This sorting order will be applied to all other tables, unless otherwise specified.
- All TEAEs by primary SOC, PT and Maximal CTCAE grade, showing number (%) of patients with at least one TEAE, sorted by SOC and PT in alphabetic order. This sorting order will be applied to all other tables, unless otherwise specified.
- All TEAEs \(\geq\) Grade 3 by primary SOC, PT and Maximal CTCAE grade
- All related TEAEs by primary SOC, PT and Maximal CTCAE grade (including possibly related, probably related, or related)
- All TEAEs leading to treatment withdrawal by primary SOC, PT and Maximal CTCAE grade
- All TEAEs leading to dose delay by primary SOC, PT and Maximal CTCAE grade
- All TEAEs leading to dose reduction by primary SOC, PT and Maximal CTCAE grade

ADCT-402-101 SAP version 1.0

All TEAEs leading to infusion interruption by primary SOC, PT and Maximal CTCAE grade

- All TEAEs with fatal outcome by primary SOC, PT and Maximal CTCAE grade
- All Serious TEAEs by primary SOC, PT and Maximal CTCAE grade
- All infusion related reaction TEAEs by primary SOC, PT and Maximal CTCAE grade
- Summary of grouped TEAEs selected by Standardised MedDRA Query (SMQ), ADCT modified SMQ will also be provided by primary Grouped term, PT and Maximal CTCAE grade. These group terms include: for effusion/edema, hepatic, fatigue, skin/nail, pain.
- Summary of TEAEs will also be provided by demographic factors including: sex, age group, race, disease subtype if appropriate.

All TEAEs, all serious adverse events (SAEs), all TEAEs leading to treatment withdrawal, all TEAEs leading to dose reduction, all TEAEs leading to dose delay, all TEAEs considered infusion related reactions, all TEAEs with fatal outcome and non-TEAEs will be listed.

#### 4.8.2.2 Deaths

The following deaths summaries will be generated on the safety analysis set.

- Number (%) of patients who died during the study and reasons for death
- Number (%) of patients who died within 30 days after last dose of study drug except deaths occurred after taking any subsequent anticancer therapy/procedure and reasons for death

All deaths will be listed.

# 4.8.3 Laboratory Data

Laboratory data of hematology, biochemistry, coagulation, and additional renal function studies up to 84 days after last dose of study drug or the end of treatment visit date, whichever is later, will be reported in SI units. Descriptive statistics (mean, standard deviation, median, and range) will be calculated for the raw data and for their changes from baseline at each scheduled assessment.

All results will be summarized using shift from baseline. Shifts for clinical laboratory results that can be graded according to CTCAE version 4.0 will be summarized by CTCAE grade.

Summaries by visit will include data from scheduled assessments, and all data will be reported according to the nominal visit date for which it was recorded. Unscheduled data will be included in "worst case post-baseline" summaries, which will capture a worst case across all scheduled and unscheduled visits after the first dose of study treatment.

Summary analyses will include data up to the start of subsequent anticancer therapy/procedure.

All laboratory data, including urinalysis, will be listed. Pregnancy test results will not be listed, but will be included in datasets.

ADCT-402
ADCT-402-101
SAP version 1.0

## 4.8.4 Electrocardiogram

Electrocardiogram (ECG) parameters (e.g., QTc in ms) will not be converted or derived, but will be reported as provided by investigational sites.

Descriptive statistics (mean, standard deviation, median, and range) will be calculated for the raw data and for their changes from baseline at each scheduled assessment.

The following abnormal QTc (including QTcF, QTcB and QTc with unspecified method) will be reported:

At any post-baseline with absolute value

```
>450 - <=480 ms
>480 - <=500 ms
> 500 ms
```

Change from Baseline

>30 - <=60 ms

>60 ms

For patients with unspecified QTc method at either baseline or post-baseline, consistent correction method is assumed within a patient when calculating the change from baseline.

Summary analyses will include data up to the start of subsequent anticancer therapy/procedure.

All ECG data will be listed, both for quantitative data and for overall impression.

## 4.8.5 Vital Signs

Descriptive statistics (mean, standard deviation, median, and range) for vital signs data, including systolic and diastolic blood pressure, heart rate, respiration rate, and body temperature will be calculated for the raw data and for their changes from baseline at each scheduled assessment.

Summary analyses will include data up to the start of subsequent anticancer therapy/procedure.

All vital signs data will be listed together with body weight and ECOG performance score.

#### 4.8.6 ECOG Performance Status

ECOG performance score data will be listed together with vital signs and body weight.

## 4.8.7 Physical Examinations and Body Weight

Physical examination will be performed according to protocol. Clinically significant findings from the physical examinations will be recorded as medical history (prior to first administration of ADCT-402) or AEs (subsequent to first administration of ADCT-402).

Body weight will be listed together with vital signs and ECOG performance score.

## 4.9 Efficacy Analyses

Disease assessment will be performed according to protocol. The endpoints described in this section use the investigator's evaluation according to the Lugano Classification criteria and clinical progression from End of Treatment (EOT)/Study disposition page.

Lesion assessment data (target lesions, non-target lesions, and new lesions) will be listed. A separate listing will contain derived data for DOR, PFS, and OS.

## 4.9.1 Overall Response Rate

Overall response rate is defined as the proportion of patients who achieve either CR or PR as best overall response as assessed by investigators according to the Lugano Classification criteria before the start of subsequent anticancer therapy or procedure.

The order of overall response category is: CR, PR, SD, NE, PD (including disease recurrence/relapse). The overall response category will be derived based on response assessment performed on or before the start of subsequent anticancer therapy/procedure. Patients without documented subsequent anticancer therapy and/or with missing start date of anticancer therapy will be considered as not having received subsequent anticancer therapy. If a patient only has one valid disease assessment which is SD, and the assessment is within 35 days after the first dose, the overall response for this patient will be considered as NE.

The overall response rate and the corresponding 95% two-sided exact confidence interval at each dose level will be presented. Subgroup analysis may be provided for disease subtype, disease stage, double/triple hit (yes/no), bulky disease (yes/no), age group, sex, country, response to the first line and/or most recent line of prior systematic therapy (relapse: CR+PR vs. refractory: SD+PD vs. other: NE + missing), and other relevant variables.

Percent change from baseline in the sum of product of diameters (SPD) for target lesions will be presented for available data in the efficacy analysis set by dose level. These data will also be displayed as a waterfall plot, with vertical bars representing the sorted values of best percent reduction for each patient.

Tumor response and lesion measurement will be listed by assessment visit.

# 4.9.2 Duration of Response

Duration of response will be defined for patients with CR or PR only as the interval between the date of initial documentation of a response and the date of first documented evidence of progressive disease (based on radiographic or clinical progression at EOT/end of study [EOS]) or death. Patients who had the event after the start of subsequent anticancer therapy/procedure, or are progression-free and alive at the time of clinical cut-off, or have unknown status, will be censored at the last valid tumor assessment on or before the start of subsequent anticancer therapy/procedure or clinical cut-off time. When a subsequent anticancer therapy is used and progressive disease (based on radiographic or clinical progression at EOT/EOS) is observed within 6 days, they will be considered as the same visit (within the +/-6 days visit window) and the patient will be counted as having an event (losing the response).

ADCT-402-101 SAP version 1.0

Duration of response will be estimated and displayed by dose levels for the efficacy analysis set using Kaplan-Meier methods (SAS® PROC LIFETEST). A Kaplan-Meier plot will be presented.

Subgroup analyses may be provided for disease subtype, disease stage, double/triple hit (yes/no), bulky disease (yes/no), age group, response to the first line and/or most recent line of prior systematic therapy (relapse: CR+PR vs. refractory: SD+PD vs. other: NE + missing), best response to ADCT-402 (CR/PR), and other relevant variables.

## 4.9.3 Time to Response:

Time to response (TTR) for the subset of patients who achieve a CR or PR will be summarized using descriptive statistics.

## 4.9.4 Progression-free Survival

Progression-free survival is defined as the interval between the date of first dose and the date of disease progression (based on radiographic or clinical progression at EOT/EOS) or death, whichever occurs first. Patients who have the event after the start of subsequent anticancer therapy/procedure, or who are progression-free and alive at the time of clinical cutoff, or have unknown status, will be censored at the time of their last valid disease assessment on or before the start of subsequent anticancer therapy/procedure or clinical cut-off. When a subsequent anticancer therapy was used and progressive disease (based on radiographic or clinical progression at EOT/EOS) were observed within 6 days, they will be considered as the same visit (within the +/-6 days window) and the patient will be counted as having an event.

Patients with no post-baseline disease assessment will be censored on Day 1.

PFS will be estimated and displayed by dose levels for the efficacy analysis set using Kaplan-Meier methods (SAS® PROC LIFETEST). Patients who do not have a PFS event during or after the study will be censored. A Kaplan-Meier plot will be presented.

#### 4.9.5 Overall Survival

Overall survival is defined as the interval between the date of first dose and the date of death from any cause. Patients who are known to be alive as of their last known status will be censored at their date of last contact. Patients who are lost to follow-up will be censored at the date the patient is last known to have been alive. The last confirmed alive date is the latest of the following: study visit date, telephone contact date, end of study last confirmed alive date, follow-up systemic (anticancer) therapy end date or start date (if ongoing or end date is missing), local or central radiologist scan date, or other date in the clinical database.

OS will be estimated and displayed by dose levels for the efficacy analysis set using Kaplan-Meier methods (SAS® PROC LIFETEST). A Kaplan-Meier plot will be presented.

## 4.10 Pharmacokinetic/Pharmacodynamics Analyses

#### 4.10.1 PK Analysis Method

The actual blood sampling time and actual amount of dose administered will be recorded and used in calculation of PK parameters. All PK samples will be evaluable as long as the actual collection times are recorded. Analysis of the ADCT-402 total antibody [drug-to-antibody ratio (DAR $\geq$ 0)], PBD-conjugated antibody (DAR $\geq$ 1), and SG3199 (unconjugated warhead) concentrations in serum were analyzed using a noncompartmental (NCA) analysis method. The PK parameters from analysis included maximum concentration (C<sub>max</sub>), time to C<sub>max</sub> (T<sub>max</sub>), area under the concentration-time curve from time zero to the last quantifiable concentration (AUC<sub>last</sub>), area under the concentration-time curve (AUC) from time zero to the end of the dosing interval (AUC<sub>tau</sub>), area under the concentration-time curve from time zero to infinity (AUC<sub>inf</sub>), accumulation index (AI), terminal half-life (T<sub>half</sub>), systemic clearance (CL), clearance (CL<sub>ss</sub>) and volume of distribution at steady state (V<sub>ss</sub>).

Data presentation by tables will include individual patient concentrations by actual time, individual PK parameters, statistical summaries for concentrations by dose cohort and nominal time, and statistical summary for PK parameters. Data presentation by figures will include individual patient concentrations by actual time, and mean (standard error) of concentrations by nominal time.

At selected times as indicated in the schedule of events tables, samples for ADCT-402 antidrug antibodies (ADA) were also collected concurrently with the PK samples. Results from ADA testing will include tabular summarization for number/proportion of patients with positive predose ADA response, number of patients with post-dose ADA response only, and number of patients with positive ADA response at any time. The denominator will be the total number of patients tested for ADAs in the study. For instances in which a positive ADA titer is observed, results from testing for neutralizing antibody potential will be considered.

| _ |
|---|

ADCT-402-101 SAP version 1.0

The results of all peripheral white blood cell populations, DNA cross-link formation, and renal functional tests will be listed by patient.

# **5 Interim Analyses**

No formal interim analysis is planned.

# 6 Data handling conventions

#### **6.1 General conventions**

## 6.1.1 Missing data

#### Handling of missing/partial dates

In general, imputation of missing dates will be made for AE onset date, AE resolution date, date of death, medication start/end dates, start and end dates of prior and subsequent therapies, and date of initial diagnosis for reporting. No imputation should be done at the data level.

- If dates are completely missing, no imputation will be made.
- For any partial date with missing year, no imputation will be made.
- For missing initial diagnosis date and subsequent therapies, if only day is missing, then the 15th of the month will be used; if only year is present, then June 30th will be used. If such imputed date for initial diagnosis is on or after date of first dose, then date of first dose 1 will be used. If such imputed date for subsequent therapies is before date of last dose, then date of last dose +1 will be used.
- If the imputed date is for an AE start date and is in the same year and month as but before the first dose date, then the first dose date will be used, or if the imputed AE start date is after the AE end date, then the AE end date will be used. If the imputed date is for an AE start date and is in the same year and month as but after the last dose date + 84 days, then the last dose date + 84 days will be used.
- If a medication date or time is missing or partially missing, so it cannot be determined whether it was taken prior or concomitantly, it will be considered as a prior and concomitant medication.
- If the imputed date is for a date of death and is before the last date that the patient is known to be alive, the latter date will be used.

#### Handling of missing relationship to investigational product of TEAEs

If the assessment of the relationship to investigational product is missing, then the relationship to investigational product has to be assumed and the TEAE considered as such in the frequency tables of possibly related TEAEs, but no imputation should be done at the data level.

#### Handling of missing severity/grades of AEs

If the severity/grade is missing for one of the treatment emergent occurrences of an AE, the maximal severity of the remaining occurrences will be considered. If the severity is missing for all the occurrences a "missing" category will be added in summary table.

No other imputation of values for missing data will be performed.

#### **6.1.2** Unscheduled visits

Unscheduled visit measurements of laboratory data, vital signs, and ECG will be used for computation of baseline and worst values and/or grades. Re-windowing for unscheduled visits will not be performed

## **6.1.3 Duplicated visits**

Depending on the statistical analysis method, single values may be required for each analysis window. For example, change from baseline by visit usually requires a single value per visit. Unless otherwise noted throughout the rest of this document, when a single value is needed, the following rule(s) will be used:

- If more than 1 assessment occurs during the same nominal visit, select the record closest to the nominal day for that visit.
- If there are 2 assessments that are equidistant from the nominal day, the data of the assessment after the scheduled study day will be used.
- The last measurement will be used if multiple measurements are taken on the same day.

# **Appendix 1 Glossary of Abbreviations**

| Glossary of Abbreviations: | |
|---|---|
| ADA | Anti-drug antibody |
| AE | Adverse event |
| AI | Accumulation index |
| AUC | Area under the concentration-time curve |
| B-NHL | B-cell lineage non-Hodgkin lymphoma |
| CBC | Complete blood count |
| CD | Cluster of differentiation |
| CI | Confidence interval |
| CL | Clearance |
| Cmax | Maximum concentration |
| CR | Complete response |
| CRF | Case report form |
| CSR | Clinical study report |
| CTCAE | Common Terminology Criteria for Adverse Events |
| DAR | Drug-to-antibody ratio |
| DESC | Dose Escalation Steering Committee |
| DLT | Dose-limiting toxicity |
| DOR | Duration of response |
| ECG | Electrocardiogram |
| ECOG | Eastern Cooperative Oncology Group |
| EOS | End of study |
| ЕОТ | End of treatment |
| IP | Investigational product |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MTD | Maximum tolerated dose |
| NCA | Noncompartmental |
| NE | Not evaluable |
| NHL | Non-Hodgkin lymphoma |
| ORR | Overall response rate |

ADCT-402-101 SAP version 1.0

| OS | Overall survival |
|------------------------|-------------------------------------------|
| PBD | Pyrrolobenzodiazepine |
| PD | Pharmacodynamics, progressive disease |
| PFS | Progression-free survival |
| PK | Pharmacokinetic |
| PR | Partial response |
| PT | Preferred term |
| Q6W | Every 6 weeks |
| QTc | Corrected QT interval (ms) |
| SAE | Serious adverse event |
| SAP | Statistical analysis plan |
| SD | Stable disease |
| SMQ | Standardised MedDRA Query |
| SOC | System organ class |
| SPD | Sum of product of diameters |
| std | Standard deviation |
| TEAE | Treatment-emergent adverse event |
| TFLs | Tables, figures, and listings |
| TTR | Time to response |
| $\Lambda_{\mathbf{z}}$ | Terminal elimination phase rate constant |
| Tmax | Time to maximum concentration |
| t <sub>1/2</sub> | Terminal half-life |
| V <sub>ss</sub> | Volume of distribution at steady-state |
| $V_z$ | Volume of distribution |
| WBC | White blood cells |
| WHO-DD | World Health Organization-Drug Dictionary |